CLINICAL TRIAL: NCT00874874
Title: Phase II Multicenter Stratified Study Evaluating the Efficacy and Toxicity of Sorafenib in Treating Locally Advanced or Metastatic Angiosarcomas That Are Not Accessible to Curative Surgery
Brief Title: Sorafenib in Treating Patients With Angiosarcoma That is Locally Advanced, Metastatic, or Unable to Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000633547; COL-Angio-Next; BAYER-COL-Angio-Next; COL-2007-10; INCA-RECF0636; EUDRACT-2007-004651-10
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-07

CONDITIONS: Sarcoma
Keywords: stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; adult angiosarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma | interventions — Sorafenib

INTERVENTIONS:
Drug: sorafenib tosylate

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sorafenib works in treating patients with angiosarcoma that is locally advanced, metastatic, or unable to be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of non-progression at 9 months in patients with unresectable, locally advanced, or metastatic angiosarcoma treated with sorafenib tosylate.

Secondary

* Determine the rate of non-progression at 60, 120, and 180 days.
* Determine the median time to progression.
* Determine overall survival.
* Determine the best response rate.
* Determine the clinical and biological factors that predict clinical benefit.
* Evaluate tolerability by NCI CTCAE v3.0.
* Correlate efficacy with plasma expression of genes implicated in controlling angiogenesis.
* Explore the tumor expression of these genes in tissue from a tumor bank.

OUTLINE: This is a multicenter study.

Patients are stratified according to disease type (cutaneous angiosarcoma [scalp, breast, or soft tissue] vs visceral angiosarcoma). All patients receive oral sorafenib tosylate twice daily for 9 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed angiosarcoma

  * Locally advanced or metastatic disease
  * Unresectable disease
* No Kaposi sarcoma, hemangiopericytoma, or hemangioendothelioma
* Measurable tumor with at least 1 measurable lesion by RECIST criteria
* Tumor in a previously irradiated area must not show progression
* No brain metastases or meningeal tumors (symptomatic or asymptomatic)

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 3 months
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* PT or INR and aPTT ≤ 1.5 times upper limit of normal (ULN)

  * Anticoagulation treatment with heparin or vitamin K allowed if the above criteria are met
* Liver transaminases ≤ 2.5 times ULN (≤ 5 times ULN in the presence of liver metastases)
* Total bilirubin ≤ 1.5 times ULN
* Serum creatinine ≤ 1.5 times ULN
* Amylase and lipase ≤ 1.5 times ULN
* Not pregnant or nursing
* Weight loss from pre-disease weight < 20% over the past 12 months
* Able to swallow
* No active or ischemic coronary artery disease
* No myocardial infarction within the past 6 months
* No NYHA class III-IV cardiac failure
* No uncontrolled hypertension
* No coagulopathy
* No active uncontrolled peptic ulcer
* No patients on renal dialysis
* No active bacterial or fungal infection > CTCAE v3.0 grade 2
* No HIV or hepatitis B or C positivity
* No chronic unstable illness that could jeopardize patient safety or compliance
* No other progressive or malignant tumor
* No known or suspected allergy to sorafenib tosylate
* No psychological, familial, social, or geographic situations that preclude clinical follow up
* No patients deprived of liberty or under guardianship
* No cardiac arrhythmia requiring antiarrhythmic medication (except beta-blockers or digoxin for chronic atrial fibrillation)
* No epilepsy requiring antiepileptic drugs

PRIOR CONCURRENT THERAPY:

* See Patient Characteristics
* No prior organ or peripheral stem cell transplantation
* No more than 2 prior lines of chemotherapy
* At least 28 days since prior treatment (systemic or major surgery)
* No concurrent therapy for another malignancy
* No concurrent CYP3A inducers (e.g., rifampicin, St. John wort, phenytoin, carbamazepine, phenobarbital, dexamethasone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Rate of non-progression at 9 months by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Penel, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

REFERENCES:
- [Derived] Penel N, Ray-Coquard I, Bal-Mahieu C, Chevreau C, Le Cesne A, Italiano A, Bompas E, Clisant S, Baldeyrou B, Lansiaux A, Robin YM, Bay JO, Piperno-Neumann S, Blay JY, Fournier C. Low level of baseline circulating VEGF-A is associated with better outcome in patients with vascular sarcomas receiving sorafenib: an ancillary study from a phase II trial. Target Oncol. 2014 Sep;9(3):273-7. doi: 10.1007/s11523-013-0299-0. Epub 2013 Nov 12. PMID 24218035
- [Derived] Valentin T, Fournier C, Penel N, Bompas E, Chaigneau L, Isambert N, Chevreau C. Sorafenib in patients with progressive malignant solitary fibrous tumors: a subgroup analysis from a phase II study of the French Sarcoma Group (GSF/GETO). Invest New Drugs. 2013 Dec;31(6):1626-7. doi: 10.1007/s10637-013-0023-z. Epub 2013 Sep 5. PMID 24005614
- [Derived] Ray-Coquard I, Italiano A, Bompas E, Le Cesne A, Robin YM, Chevreau C, Bay JO, Bousquet G, Piperno-Neumann S, Isambert N, Lemaitre L, Fournier C, Gauthier E, Collard O, Cupissol D, Clisant S, Blay JY, Penel N; French Sarcoma Group (GSF/GETO). Sorafenib for patients with advanced angiosarcoma: a phase II Trial from the French Sarcoma Group (GSF/GETO). Oncologist. 2012;17(2):260-6. doi: 10.1634/theoncologist.2011-0237. Epub 2012 Jan 27. PMID 22285963